CLINICAL TRIAL: NCT06689384
Title: The Effect of "Cut-out-Rescan" Procedure Under Rubber-Dam Isolation on the Trueness of Intraoral Scanners
Brief Title: Cut-out-Rescan Procedure Under Rubber-Dam Isolation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2024.1000
Record Dates: First submitted 2024-11-08; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Trueness; Intraoral Scanner; Rubberdam
Keywords: Trueness; intraoral scanner; cut-out-rescan; rubberdam; indirect restoration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Recording of the diagnostic 3D images (Experimental): 20 patients with adequate oral health who had daily routine appointments for treatment at Marmara University restorative dentistry department were included in the study. Exclusion criteria for the study were missing premolar and molar teeth (except wisdom teeth) or the presence of amalgam and ceramic restorations that could affect the scanning in the right hemi-arc of the mandible. Using of intra oral scanners was performed by a restorative dentist with 5 years of experience. were scanned with 4 different intraoral scanners (IOS) (Trios 3, 3Shape; Primescan, Dentsply; Element 5D, iTero; Lumina, iTero) prior to the procedure, and the obtained digital impressions were stored as a standard tessellation language (STL) file. The digital scan had appropriate anatomic references to enable a proper matching with the digital scan taken after teeth preparation. The official scanning strategy and ambient scanning light conditions in the manufacturer's instructions were followed for all scanners.
  Interventions: Device: Taking images from the right lower jaw with an intraoral scanner
- Rubberdam Isolation (Experimental): The 2nd premolar, 1st, and 2nd molar teeth were isolated with a rubber dam (medium; Nic Tone, Manufacturera Dental Continental) to be included in the operation field. Clamps were placed on the 2nd premolar and 2nd molar teeth. It was aimed to facilitate the second scanning process by expanding the isolation area to include 3 teeth. A flowable composite was applied by placing Teflon tape on the occlusal surface of the 1st molar to create a difference in its morphology. In the procedure that simulated the final impression process under rubber dam isolation, the relevant tooth was marked on the initial scan along with the contact areas of the adjacent teeth. The marked area which the to be re-scanned, was trimmed away from the virtual casts. The diameter of the mesh holes was controlled by adjusting the settings of the automatic mesh hole generator in the software program of the IOS.
  Interventions: Procedure: Clamp placement on canine and 2nd molar teeth and rubberdam rubber band insertion
- Selective Cutting on the Scanner (Experimental): In the procedure that simulated the final impression process under rubber dam isolation, the relevant tooth was marked on the initial scan along with the contact areas of the adjacent teeth. The marked area which the to be re-scanned, was trimmed away from the virtual casts. The diameter of the mesh holes was controlled by adjusting the settings of the automatic mesh hole generator in the software program of the IOS.
  Interventions: Device: Taking images from the right lower jaw with an intraoral scanner
- Recording the Final 3D Image (Experimental): Subsequently, the mesh hole area was rescanned starting on the occlusal surface of the second molar, moving toward the occlusal of the first molar to the occlusal of the second premolar, then the buccal surfaces of the second premolar, followed by the first molar and second molar. The rescanning procedures ended with the lingual surfaces of the second molar, followed by the lingual surfaces of the first molar and second premolar. Following the second scan, the area was re-scanned in high-resolution mode, where higher mesh quality could be achieved. The software of the intraoral scanner automatically fused two different data sets obtained by initial/reference and preparation digital scans. Data about tooth positions, morphologies, rubber dam, and surrounding soft tissues was integrated simultaneously. The obtained final scan was exported as an STL file.
  Interventions: Device: Taking images from the right lower jaw with an intraoral scanner

INTERVENTIONS:
Device: Taking images from the right lower jaw with an intraoral scanner — The patients' mandibular arches were scanned with 4 different intraoral scanners (IOS) (Trios 3, 3Shape; Primescan, Dentsply; Element 5D, iTero; Lumina, iTero) prior to the procedure, and the obtained digital impressions were stored as a standard tessellation language (STL) file. The 2nd premolar, 1st, and 2nd molar teeth were isolated with a rubber dam (medium; Nic Tone, Manufacturera Dental Continental) to be included in the operation field. Clamps were placed on the 2nd premolar and 2nd molar teeth. Subsequently, the mesh hole area was rescanned starting on the occlusal surface of the second molar, moving toward the occlusal of the first molar to the occlusal of the second premolar, then the buccal surfaces of the second premolar, followed by the first molar and second molar.
  Arms: Recording of the diagnostic 3D images; Recording the Final 3D Image; Selective Cutting on the Scanner
Procedure: Clamp placement on canine and 2nd molar teeth and rubberdam rubber band insertion — The 2nd premolar, 1st, and 2nd molar teeth were isolated with a rubber dam (medium; Nic Tone, Manufacturera Dental Continental) to be included in the operation field. Clamps were placed on the 2nd premolar and 2nd molar teeth. It was aimed to facilitate the second scanning process by expanding the isolation area to include 3 teeth.
  A flowable composite was applied by placing Teflon tape on the occlusal surface of the 1st molar to create a difference in its morphology.
  Arms: Rubberdam Isolation

SUMMARY:
Aim: This clinical study investigated the effect of the "cut-out-rescan" procedure under rubber dam isolation on restorative scanning trueness of four intraoral scanners.

Materials and Methods: The initial scans were collected from 20 patients using 4 dental intraoral scanners (Trios 3, 3Shape; Cerec Primescan, Dentsply Sirona; iTero Element 5D, Align; iTero Lumina, Align). The 3-dimensional data was obtained from the right or left side of the mandibula between the canine-to-2nd molar area and recorded in .stl format. Then the 2nd premolar was cut with the cutting tool in the related scanner software in a range including 1mm from the adjacent teeth. The determined area was clinically isolated with the rubber-dam and the same quadrant was rescanned to let the software overlap with the cut-out area. The overlapped scan was recorded in .stl format as the second scan data. The first and second scan data from the 4 scanners were then transferred to the Oracheck (Dentsply Sirona) software program and digitally overlapped to measure the conformity. The deviations detected in the 1st premolar, 2nd premolar, and 1st molar were selectively and jointly assessed in distance (mm) and volume (mm3) for every scanner data. Robust ANOVA and Kruskal Wallis tests were used for the statistical analyses and the significance level was set at <.050.

DETAILED DESCRIPTION:
The CAD/CAM system has been in use in the industry for decades and has been popular in recent years with its use in many areas of dentistry. These systems' numerous advantages over conventional methods, coupled with the ongoing advancement of intraoral scanner technologies, have led to their frequent preference among clinicians. It is well known that the method of rescanning, which is frequently employed in clinical settings to acquire data from previous, can also affect the accuracy of the results. In addition, it has been observed that the efficacy of the rescanning method varies depending on the intraoral scanner utilized.. On the other hand, the "cut-out-rescan" technique is a procedure performed on a prepared tooth that involves cutting and rescanning the tooth based on a previously performed diagnostic scan.Considering this information, the objective of this in vivo study was to assess the accuracy of four different scanners using a cut-out-rescan procedure with a rubber dam isolation. This clinical study was conducted with the approval of a local ethics committee (Protocol number: 09.2024.1000). Informed consent was obtained from each patient. 20 patients with adequate oral health who had daily routine appointments for treatment at Marmara University restorative dentistry department were included in the study. Exclusion criteria for the study were missing premolar and molar teeth (except wisdom teeth) or the presence of amalgam and ceramic restorations that could affect the scanning in the right hemi-arc of the mandible. Using of intra oral scanners was performed by a restorative dentist with 5 years of experience.The patients' mandibular arches were scanned with 4 different intraoral scanners (IOS) (Trios 3, 3Shape; Primescan, Dentsply; Element 5D, iTero; Lumina, iTero) prior to the procedure, and the obtained digital impressions were stored as a standard tessellation language (STL) file. The digital scan had appropriate anatomic references to enable a proper matching with the digital scan taken after teeth preparation. The official scanning strategy and ambient scanning light conditions in the manufacturer's instructions were followed for all scanners. A 15-minute break was taken between the different experimental groups to reduce operator fatigue, and the IOS was calibrated before each experimental scan according to the manufacturer's recommendations.The 2nd premolar, 1st, and 2nd molar teeth were isolated with a rubber dam (medium; Nic Tone, Manufacturera Dental Continental) to be included in the operation field. Clamps were placed on the 2nd premolar and 2nd molar teeth. It was aimed to facilitate the second scanning process by expanding the isolation area to include 3 teeth.

A flowable composite was applied by placing Teflon tape on the occlusal surface of the 1st molar to create a difference in its morphology. In the procedure that simulated the final impression process under rubber dam isolation, the relevant tooth was marked on the initial scan along with the contact areas of the adjacent teeth. The marked area which the to be re-scanned, was trimmed away from the virtual casts. The diameter of the mesh holes was controlled by adjusting the settings of the automatic mesh hole generator in the software program of the IOS. Subsequently, the mesh hole area was rescanned starting on the occlusal surface of the second molar, moving toward the occlusal of the first molar to the occlusal of the second premolar, then the buccal surfaces of the second premolar, followed by the first molar and second molar. The rescanning procedures ended with the lingual surfaces of the second molar, followed by the lingual surfaces of the first molar and second premolar. Following the second scan, the area was re-scanned in high-resolution mode, where higher mesh quality could be achieved. The software of the intraoral scanner automatically fused two different data sets obtained by initial/reference and preparation digital scans. Data about tooth positions, morphologies, rubber dam, and surrounding soft tissues was integrated simultaneously. The obtained final scan was exported as an STL file. The discrepancy examination was achieved using the Oracheck Software (Dentsply Sirona, Germany) program, which allows for a 3D comparison between two digital scans utilizing the best-fit algorithm. The initial/reference and final STL files were imported into the software program and three-dimensional images of the 2nd premolar, 1st molar and 2nd molar teeth were superimposed. Gingiva and rubber dam records were removed from the digital models with the "cutting" and "editing" tools. Deviations between models were obtained and recorded volumetric (mm3) and distance (mm) and analyzed quantitatively. Trueness was defined as the average absolute distance between the initial and the final digital scans.Data were analysed with IBM SPSS v23 and Jamovi software. The conformity of the data to normal distribution was analysed by Shapiro-Wilk test. Since the data by tooth and scanner were not normally distributed, they were analysed by Robust ANOVA using the WALRUS package. Intraoral general evaluations were analysed by Kruskal Wallis test. Multiple comparisons were made with Bonferroni Test. The relationship between quantitative data that did not show normal distribution was analysed by Spearman's rho correlation. Intraobserver agreement was analyzed with intraclass correlation coefficient. Median (minimum-maximum) was used to represent quantitative data. Significance level was taken as p<0.050.

ELIGIBILITY:
Inclusion Criteria:

* l8-65 age range
* Have sufficient cognitive ability to understand the consent procedure
* To have clinically healthy gingiva and periodontium
* Daily cigarette consumption of 10 cigarettes or less
* No loss of attachment, bleeding or plaque accumulation on probing
* Vital mandibular teeth without signs of irreversible pulpitis
* Caries in the right or left lower 2nd premolar tooth suitable for direct composite restoration indication
* The 1st molar, 2nd molar, 1st premolar and canine teeth in the relevant region are not missing and do not contain any fixed prosthesis

Exclusion Criteria:

* Any disability (mental health conditions, mental disabilities and physical disabilities)
* Systemic diseases or medically serious risks (cardiovascular disorder, diabetes, hypertensive, epileptic)
* Gingival hyperplasia or periodontal disease
* Symptoms of periapical or pulpal pathology
* Non-vital endodontically treated teeth
* Teeth showing mobility
* Congenital tooth deficiencies
* Having a prominent crossbite, missing teeth, jaw anomaly or prosthetic restoration in the relevant region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Recording diagnostic 3D- image with Trios 3 intraoral scanner | Up to 5 days
  The diagnostic (first) 3D images were taken with Trios 3 from the right mandible of the patients. With the camera-containing tip of the intraoral scanner, the 3D image of the patient's right mandible was saved in the scanner's memory and can be examined in 3D in STL format on the computer screen. The scanners record multiple photographs while travelling through the patient's mouth with the camera and automatically combine them with the software to obtain a three-dimensional image.
Recording diagnostic 3D-image with Primescan intraoral scanner | up to 5 days
  The diagnostic (first) 3D images were taken with Primescan from the right mandible of the patients. With the camera-containing tip of the intraoral scanner, the 3D image of the patient's right mandible was saved in the scanner's memory and can be examined in 3D in STL format on the computer screen. The scanners record multiple photographs while travelling through the patient's mouth with the camera and automatically combine them with the software to obtain a three-dimensional image
Recording diagnostic 3D-image with Itero Element 5D intraoral scanner | up to 5 days
  The diagnostic (first) 3D images were taken with Element 5D from the right mandible of the patients. With the camera-containing tip of the intraoral scanner, the 3D image of the patient's right mandible was saved in the scanner's memory and can be examined in 3D in STL format on the computer screen. The scanners record multiple photographs while travelling through the patient's mouth with the camera and automatically combine them with the software to obtain a three-dimensional image.
Recording diagnostic 3D-image with Lumina intraoral scanner | up to 5 days
  he diagnostic (first) 3D images were taken with Lumina from the right mandible of the patients. With the camera-containing tip of the intraoral scanner, the 3D image of the patient's right mandible was saved in the scanner's memory and can be examined in 3D in STL format on the computer screen. The scanners record multiple photographs while travelling through the patient's mouth with the camera and automatically combine them with the software to obtain a three-dimensional image
Applying rubberdam isolation to patients | up to 5 days
  On the 3rd and 7th teeth, rubber dam isolation was applied by placing a clamp. Threads were not involved during retraction. Only the gums were covered with rubber dam rubber and the teeth remained exposed.
Selective cutting from image on Trios 3 intraoral scanner | up to 5 days
  Using the computer software of the Trios 3 intraoral scanner and editing the screen of the scanner, the entire tooth number 5 in the 3D image and 1 mm of the adjacent teeth 4 and 6 were cut out.
Selective cutting from image on Primescan intraoral scanner | up to 5 days
  Using the computer software of the Primescan intraoral scanner and editing the screen of the scanner, the entire tooth number 5 in the 3D image and 1 mm of the adjacent teeth 4 and 6 were cut out
Selective cutting from image on Itero Element 5D intraoral scanner | up to 5 days
  Using the computer software of the Element 5D intraoral scanner and editing the screen of the scanner, the entire tooth number 5 in the 3D image and 1 mm of the adjacent teeth 4 and 6 were cut out
Selective cutting from image on Lumina intraoral scanner | up to 5 days
  Using the computer software of the Lumina intraoral scanner and editing the screen of the scanner, the entire tooth number 5 in the 3D image and 1 mm of the adjacent teeth 4 and 6 were cut out

SECONDARY OUTCOMES:
Recording final image with Trios 3 intraoral scanner | up to 5 days
  The selectively cut region was scanned again with Trios 3 during rubberdam isolation and the final image was obtained.The final 3D images were taken with Trios 3 from the right mandible of the patients. With the camera-containing tip of the intraoral scanner, the 3D image of the patient's right mandible was saved in the scanner's memory and can be examined in 3D in STL format on the computer screen. The scanners record multiple photographs while travelling through the patient's mouth with the camera and automatically combine them with the software to obtain a three-dimensional image.
Recording final image with Primescan intraoral scanner | up to 5 days
  The selectively cut region was scanned again with Primescan during rubberdam isolation and the final image was obtained.The final 3D images were taken with Primescan from the right mandible of the patients. With the camera-containing tip of the intraoral scanner, the 3D image of the patient's right mandible was saved in the scanner's memory and can be examined in 3D in STL format on the computer screen. The scanners record multiple photographs while travelling through the patient's mouth with the camera and automatically combine them with the software to obtain a three-dimensional image.
Recording final image with Itero Element 5D intraoral scanner | up to 5 days
  The selectively cut region was scanned again with Element 5D during rubberdam isolation and the final image was obtained.The final 3D images were taken with Element 5D from the right mandible of the patients. With the camera-containing tip of the intraoral scanner, the 3D image of the patient's right mandible was saved in the scanner's memory and can be examined in 3D in STL format on the computer screen. The scanners record multiple photographs while travelling through the patient's mouth with the camera and automatically combine them with the software to obtain a three-dimensional image.
Recording final image with Lumina intraoral scanner | up to 5 days
  The selectively cut region was scanned again with Lumina during rubberdam isolation and the final image was obtained.The final 3D images were taken with Lumina from the right mandible of the patients. With the camera-containing tip of the intraoral scanner, the 3D image of the patient's right mandible was saved in the scanner's memory and can be examined in 3D in STL format on the computer screen. The scanners record multiple photographs while travelling through the patient's mouth with the camera and automatically combine them with the software to obtain a three-dimensional image.
Registration of diagnostic and final 3D images obtained from Trios 3 scanner | Between days 5 and 10
  The two (first and final) 3D- images were transferred to the Oracheck program in STL format and the difference was recorded in terms of volume (mm3) and distance (mm). After overlapping the two images, the programme automatically displayed the differences. The differences were automatically displayed in volumetric (mm3) and distance (mm).
Registration of diagnostic and final 3D images obtained from Primescan scanner | between days 5 and 10
  The two (first and final) 3D- images were transferred to the Oracheck program in STL format and the difference was recorded in terms of volume (mm3) and distance (mm). After overlapping the two images, the programme automatically displayed the differences. The differences were automatically displayed in volumetric (mm3) and distance (mm).
Registration of diagnostic and final 3D images obtained from Itero Element 5D scanner | between days 5 and 10
  The two (first and final) 3D- images were transferred to the Oracheck program in STL format and the difference was recorded in terms of volume (mm3) and distance (mm). After overlapping the two images, the programme automatically displayed the differences. The differences were automatically displayed in volumetric (mm3) and distance (mm).
Registration of diagnostic and final 3D images obtained from Lumina scanner | between days 5 and 10
  The two (first and final) 3D- images were transferred to the Oracheck program in STL format and the difference was recorded in terms of volume (mm3) and distance (mm). After overlapping the two images, the programme automatically displayed the differences. The differences were automatically displayed in volumetric (mm3) and distance (mm).
Statistical Analysis | between days 10 and 15 (last 5 days of study)
  The differences recorded were divided into two main categories: volumetric (mm3) and distance (mm). intraoral scanners were compared with each other in terms of volumetric and distance. Differences were defined as the "deviation" of the scanners from the main image.

CONTACTS AND LOCATIONS:
Overall Officials: Bora Korkut, Associate Professor, Study Director — Marmara University; Ayse Asli Senol, Asisstant Professor, Principal Investigator — Marmara University; Cevdet Can Saygılı, Research Assistant, Principal Investigator — Marmara University; Bengü Doğu Kaya, Research Asisstant, Principal Investigator — Marmara University
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
When the study is published, it will be shared.
Supporting Information: Study Protocol, CSR